CLINICAL TRIAL: NCT01994603
Title: Preventing FAS/ARND in Russian Children/Expansion to Interdisciplinary HIV Prevention in Women
Brief Title: Expansion to Interdisciplinary HIV Prevention in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1590; 3R01AA016234-05S1 (NIH)
Record Dates: First submitted 2013-10-23; First posted 2013-11-26 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: HIV; AIDS; Fetal Alcohol Syndrome; Alcohol Related Neurodevelopmental Disorder
Keywords: Prevention; HIV; AIDS; Fetal Alcohol Syndrome (FAS); Alcohol Related Neurodevelopmental Disorder (ARND)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Fetal Alcohol Spectrum Disorders | interventions — Focus Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Opt-in testing (Experimental): Participants will be scheduled for a two-hour appointment to complete the written consent procedure, enroll in the study, and participate in the study activities, testing and a focus group. Opt-in: Common barriers to HIV screening testing will be removed as much as possible (i.e., providing rapid testing, results shortly available, testing on-site, confidentiality). "There is voluntary HIV testing available to all study participants if you wish to do it. "
  Interventions: Behavioral: Opt-in or Opt-out testing; Behavioral: Focus Group
- Opt-out testing (Experimental): Participants will be scheduled for a two-hour appointment to complete the written consent procedure, enroll in the study, and participate in the study activities, testing and a focus group. Opt-out multicomponent testing. Participants will be informed that a bundled routine health test is available on a voluntary basis to study participants, and the participant may elect to decline all or part of the testing.
  Interventions: Behavioral: Opt-in or Opt-out testing; Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Opt-in or Opt-out testing — Study participants will be offered a health screening onsite.
Behavioral: Focus Group — Study participants will be invited to participate in a focus group discussion.

SUMMARY:
This trial will pilot test intervention strategies to increase utilization of HIV testing and gain knowledge for designing a clinical trial to evaluate prevention strategies to reduce HIV sexual transmission in the general population in Russia. The study will assess whether external (cost, convenience) or internal factors (low perception of own risk, reluctance to identify a partner as at-risk, fear of stigma) drive Russian women's reluctance to be tested and if peer support impacts their decision. A randomized experimental manipulation, comparing opt-in vs. bundled opt-out testing approaches, followed by focus group discussions, followed by a second-chance testing offer will be used to inform these questions. The answers will enable the international research team to engineer and then test an HIV testing promotion strategy in Russia. The project will collect preliminary data for a larger study to develop an evidence-based program to reduce the HIV transmission in this high risk population.

DETAILED DESCRIPTION:
A mixed methods research design combining qualitative and quantitative data collection methods will be used to increase the understanding of barriers to HIV testing, identify promising strategies to increase testing, generate research hypotheses, and design a future randomized clinical trial to evaluate HIV prevention targeted to at-risk women in the general population in Russia. The qualitative methods include structured interviews and a focus group participation to assess women's reasons for being the tested and possible prevention strategies. The quantitative methods include observation/recording of women's testing behaviors.

ELIGIBILITY:
Inclusion Criteria:

* A parent study participants who completed HIV risk survey and
* Reported two or more partners in the last 12 months and no or inconsistent condom use in the last 3 months and no HIV testing in the last 12 months
* Or reported any sexually-transmitted disease and no HIV testing in the last 12 months

Exclusion Criteria:

* A parent study participants who declined to be contacted for participating in future research studies

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who completed HIV test | First 1: at initial contact, an expected average of 15 minutes
  A brief survey completed over the phone. Participants asked when the last HIV test was completed and her reasons for taking the test.
Number of participants who accepted a rapid health screening/HIV test | Phase 2: an expected average of 2 hours
  Women's decision to take/not take a health screening test/HIV test is recorded. If a woman chooses to be tested, she will be asked a few questions to assess her reasons for being tested. She will be provided with the results of the testing. If a woman's test is positive for HIV (or other health risks in the bundled opt-out condition), counseling with a trained study nurse, physician or psychologist will be available on-site and a referral for additional testing, counseling, and appropriate medical care will be provided.

SECONDARY OUTCOMES:
Brief survey to assess reasons for being tested | Phase 2: at time of completing HIV testing
  Participants who accepted a rapid health screening/HIV test are asked about reasons for taking the test at this time

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Balachova, Principal Investigator — University of Oklahoma; Alla Shaboltas, PhD, Principal Investigator — Saint Petersburg State University, Russia
Locations (2):
- University of Oklahoma, Oklahoma City, Oklahoma, United States
- St. Petersburg State University, Saint Peterburg, Russia